CLINICAL TRIAL: NCT07378982
Title: Three Dimensionally Printed Ceramic-Filled Photopolymer Resin Versus CAD/CAM Resin Composite Overlays for Restoration of Extensively Damaged Endodontically Treated Posterior Teeth. An 18-month Follow-up Randomized Controlled Trial
Brief Title: 3D Printed Ceramic-Filled Photopolymer Resin Vs. CAD/CAM Resin Composite Overlays for Restoration of Extensively Damaged Endodontically Treated Posterior Teeth. An 18-month Follow-up
Acronym: 3D CAD/CAM RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Khairy Elmorsy, PhD Candidate in Restorative & Esthetics Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cairo U, Faculty of Dentistry
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Endodontically Treated Molar; Dental Restoration, Permanent
Keywords: 3D printing; CAD/CAM milling; Overlay restoration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The Intervention Group will receive 3D-printed overlay restorations for endodontically treated molar teeth.
  Interventions: Procedure: 3D printed overlay restorations
- Control Group (Active Comparator): The Control Group will receive CAD/CAM milled overlay restorations for endodontically treated molar teeth.
  Interventions: Procedure: CAD/CAM restorations

INTERVENTIONS:
Procedure: 3D printed overlay restorations — Computer-aided design (CAD) will be done by a 3D designing software (ExoCAD), and files will be created in CAD generated model file (STL format file). Then it will be placed in a nesting software (CHITOBOX) to create a Color-dependent Plot Style Table extension file (.ctb). Placement of the restoration in the nesting software will be at 30-45 degrees to increase precision of the printed restoration. (Metin et al., 2024) Then 3D printing of the restoration using a 4K LCD printer (Microdent 1 Pro, Mogassam, Egypt).
  After Printing of the restoration, the excess resin will air dried then placed in 99 % ethanol ultrasonic bath for 5 minutes followed by air dryness to romove excess uncured resin, follwed by post-curing in a nitrogen enviroment curing box with otoflash mode (LED Curing machine N1, Inox MENA) for 180-240 seconds. (Özden and Altınok Uygun, 2025), (Lim et al., 2024)
  Other Names: additive manufacturing
  Arms: Intervention
Procedure: CAD/CAM restorations — Computer designing and machining (milling): Computer-aided design (CAD) will be done using 3D designing software (ExoCAD), an STL format file will be exported to the milling machine. Then restoration from Composite blocks will be wet milled using a 5-axis milling machine. Same steps regarding glazing and polishing will be done same to the intervention group.
  Other Names: subtractive manufacturing
  Arms: Control Group

SUMMARY:
II. Introduction:

6. Background and rationale: Restoring badly mutilated teeth was and has always been a challenge in restorative dentistry. In order to solve this issue, different approaches have been proposed, including cuspal protection or cuspal coverage. This proved to increase the fracture resistance of remaining tooth structure and overall survivability of endodontically treated teeth. Different materials and techniques have been proposed to attain cuspal coverage, such as using indirect milled or pressed ceramics, indirect milled composite, and direct composite restorations(Abu-Awwad, 2019).

The integration of 3D printing in dentistry has revolutionized the fabrication of permanent indirect restorations, including inlays, onlays, and overlays. Evaluation of whether the mechanical properties, clinical feasibility, and accuracy of 3D-printed resin restorations are compared to traditional milled and pressed alternatives. Key findings highlight superior marginal fit, cost-efficiency, and adaptability of 3D-printed resins, while addressing limitations such as stain susceptibility and long-term durability

Research question:

Does a 3D printed ceramic-filled photopolymer resin show any difference in clinical performance when compared to a CAD/CAM milled composite in restoring badly decayed endodontically treated posterior teeth?

Statement of the problem:

The problems of indirect milled composites include the initial cost of the milling machine, running cost of machine repairs, bur changes, and the cost of discs and blocks, not to mention that the concept of milling as a manufacturing process has an unavoidable loss of material. (Josic et al., 2023)

Rationale for conducting the research:

Indirect restorations, such as inlays (without cusp coverage), onlays (partial cusp coverage), and overlays (full cusp coverage), aim to preserve tooth structure while restoring function and esthetics. Historically, these restorations were fabricated using ceramics or composite resins via subtractive milling or heat-pressing techniques. However, 3D printing has emerged as a transformative technology, enabling additive manufacturing of resin-based restorations with enhanced precision and reduced material waste. (Tribst et al., 2024)

Review of literature:

Extensively destructed endodontically treated molars may represent a high-risk restorative scenario due to loss of internal dentin support and undermined cusps leading to increased flexure, stress concentration and analysis, making failure more likely to occur due to cuspal fracture, bulk fracture, tooth splitting or adhesive debonding rather than simple marginal defects. Contemporary restorative concepts therefore emphasize preserving remaining tooth structure while providing cuspal coverage through adhesively bonded partial-coverage restorations like onlays, overlays and endocrowns, aiming to redistribute occlusal loads and reduce catastrophic tooth fracture. Clinical reviews of root-filled teeth consistently highlight that prognosis depends less on "endodontic status" itself and more on the quantity and quality of remaining coronal tissue, presence of ferrule, and the capacity of the definitive restoration to protect the tooth under function.

Among current treatment options, direct resin composite restorations remain attractive for being conservative, repairable, and cost-efficient. However, the effectiveness of this treatment modality decreases as cavity size leading to increased polymerization shrinkage stresses, reduced cuspal stiffness as a result of increased cavity depth, difficulty in achieving durable proximal anatomy in very large defects, and technique sensitivity under moisture compromised isolation, which can translate into higher risk of fracture or marginal breakdown over time. Indirect restorations including full crowns, partial-coverage ceramic restorations, and resin-based CAD/CAM restorations can provide better anatomic control and cuspal coverage, but has some drawbacks like added steps, cost, and may require more tooth reduction depending on design and material used.

Systematic review and meta-analysis evidence focusing specifically on endodontically treated posterior teeth suggests that outcomes between direct composite and indirect approaches can be broadly comparable in some settings, but there is a tendency for indirect restorations to be favored as defect severity increases and remaining walls decrease, while direct restorations may be more appropriate for smaller defects; importantly, the available evidence is heterogeneous and often limited by variation in preparation design, materials, and follow-up.

DETAILED DESCRIPTION:
III. Methods

A) Participants, interventions & outcomes

9. Study settings: This clinical study will be held in the clinic of Conservative dental department-Faculty of Dentistry Cairo University, Egypt.

10. Eligibility criteria:

1. Eligibility criteria of participants:

   Inclusion criteria Exclusion criteria

   • Age: 18-60 years.
   * Males or females.
   * Participants with endodontically treated molar teeth. lower molars indicated for onlay (one or two missing cusps)
   * Patients with at least 20 teeth under occlusion.
   * Good oral hygiene.
   * Co-operative patients approving to participate in the trial.
   * Have sufficient cognitive ability to understand consent procedures. • Participants with parafunctional habits or bruxism.
   * Participants with systemic diseases or disabilities that may affect participation.
   * Heavy smoking.
   * Pregnancy.
   * Lack of compliance.
   * Severe or active periodontal disease.
   * Cognitive impairment
2. Eligibility criteria for teeth:

Inclusion criteria Exclusion criteria

• Badly destructed endodontically treated molars teeth indicated for cuspal total cuspal coverage (Overlay restoration)

* No signs or symptoms after endodontic treatment.
* No signs of clinical mobility.
* Teeth with healthy periodontium. • Periapical pathosis indicating failure in endodontic treatment.
* Vital teeth.
* Signs of pathological wear.
* Severe periodontal affection or tooth indicated for extraction.
* Signs of Vertical root fracture.

  11. Interventions
  1. Examination and diagnosis:

     Examination and selection of patients will be done according to inclusion and exclusion criteria. Personal data, medical and dental history will be recorded for each participant. Clinical examination will be done using mouth mirror, explorer, standardized photographs, and periapical digital radiographs to confirm the molar teeth have extensive tissue loss and endodontic treatments were performend correctly and the teeth are indicated for cuspal coverage. A diagnostic chart will be filled providing the previously mentioned information.

     Informed Consent: Eligible participants are informed with the procedure and an informed consent will be signed.
  2. Tooth preparation procedure for both intervention and comparator:

     After patient preparation, local anesthesia will be administered, followed by rubber dam isolation. A pear shaped burs, tapered diamond burs with rounded end and a flame burs will be used with copious amount of air-water coolant for tooth preparation. Occlusal reduction will be performed ensuring a butt joint preparation for all cusps. Occlusal clearance will be achieved by a wheel or flame stone to achieve a 2 mm clearance. Prepared tooth will be air abraided using 29 µm Aluminum Oxide (Aquacare from Velopex, England).
  3. Immediate Dentin Sealing (IDS) and Cavity Design Optimization (COD):

     Immediate dentin sealing will be performed after tooth preparation to improve bond strength to freshly cut dentin and facilitate the delivery of indirect restoration as bonding will be done to mostly a hydrophobic surface. Air dryness of the cavities for 5 seconds will be performed using the air/water syringe followed by aicd etching to dentin for 5-10 seconds to remove any aluminm oxide powder residues, then application of universal adhesive (One Coat 7 Universal, Coltene, Switzerland) over all the dentine surfaces using micro-brush following manufacturer's recommendations. The adhesive will be applied and actively rubbed for 20 seconds; followed by air-thinning for solvent evaporation. Light curing will be done using a LED light-cure device ( Elipar S10, 3M ESPE, Germany).

     A layer of flowable composite will be applied on the adhesive layer to , block undercuts, or elevate the preparation which will improve the adaptation of subsequent restorations. Following this procedure, any excess adhesive will be removed with a diamond bur to expose enamel margins rendering an improved cementation and retention of restorations.

  e) Optical impression: (Intra Oral Scanning) The overlay preparations for the indirect restorations will be scanned using a calibrated Medit I600 intraoral scanner. (Medit Co., LTD, Seoul, Korea).

  f) Temporization: The prepared cavity will be coated with a layer of glycerin to allow easy removal. A light-cured temporary restoration will be applied on the cavity, and excess material will be removed after allowing the patient to bite. Initial curing will be accomplished while the patient is biting for 10 seconds followed by additional 10 seconds curing.

  g) Fabrication of indirect restorations:
* Fabrication of intervention (3D printing):

Computer-aided design (CAD) will be done by a 3D designing software (ExoCAD), and files will be created in CAD generated model file (STL format file). Then it will be placed in a nesting software (CHITOBOX) to create a Color-dependent Plot Style Table extension file (.ctb). Placement of the restoration in the nesting software will be at 30-45 degrees to increase precision of the printed restoration. (Metin et al., 2024) Then 3D printing of the restoration using a 4K LCD printer (Microdent 1 Pro, Mogassam, Egypt).

After Printing of the restoration, the excess resin will air dried then placed in 99 % ethanol ultrasonic bath for 5 minutes followed by air dryness to romove excess uncured resin, follwed by post-curing in a nitrogen enviroment curing box with otoflash mode (LED Curing machine N1, Inox MENA) for 180-240 seconds. (Özden and Altınok Uygun, 2025), Removal of supports and finishing of sharp surfaces, then air abrasion using 50 µm Aluminum Oxide with 1-2 bar for 10 to 15 seconds, followd by ultrasonic bath in distilled water to remove any residual powder. Restorations will be dried thoroughly followed by glaze application to create very smooth but thin layer, and then repeating post-curing step for 5-10 minutes.

• Fabrication of comparator (CAD/CAM): Computer designing and machining (milling): Computer-aided design (CAD) will be done using 3D designing software (ExoCAD), an STL format file will be exported to the milling machine. Then restoration from Composite blocks will be wet milled using a 5-axis milling machine. Same steps regarding glazing and polishing will be done same to the intervention group.

h) Cementation procedure: After checking the fit of restorations, the tooth surface and Intaglio surface of the restoration will for both comparator and intervention groups will be pre-treated according to the manufacturer's instructions. 50 µm aluminum oxide using the intraoral sandblaster unit followed by distilled water ultrasonic bath for removal of any residual powder, then silane coupling agent for 1 minute followed by air dryness.

Surface treatment of the tooth: After rubber dam isolation, the tooth surface will be cleaned by 50 µm aluminum oxide using the intraoral sandblaster unit. Acid etching of prepared tooth with 37% phosphoric acid for 30 seconds followed by rinsing for 30 seconds and air dryness.

i) The bonding procedure: Universal adhesive will be applied according to the manufacturer's instructions and won't be light cured until the cement application "Co-curing". Injectable resin composite will be used for the cementation of both intervention and comparator groups. Injectable composite will be placed into the prepared tooth, followed by application and proper seating of the restorations. Before light curing, proximal contact will be checked, and excess material will be removed with dental floss. After curing, occlusion will be checked and adjusted. Finishing and polishing will follow using yellow coded tapered diamond stones and Polishing using rubber points mounted on a low-speed handpiece.

12. Outcomes: Clinical assessment using Modified USPHS criteria 14. Sample size: Sample size was calculated based on the primary outcome used in the reference trial (modified USPHS categorical rating, dichotomized as clinically ideal "Alpha" versus non-ideal scores), and assuming the same expected distribution between groups. With a two-sided α error of 0.05 and 80% power, the anticipated proportions were 0.99 Alpha and 0.01 non-Alpha for the CAD/CAM milled composite group and 0.85 Alpha and 0.15 non-Alpha for the 3D-printed ceramic-filled photopolymer resin group, corresponding to a large effect size (w = 0.7) using a Chi-square test. The minimum required sample was 26 restorations; to compensate for an anticipated 20% attrition rate, the final sample size was increased to 32 restorations (16 restorations per group). Sample size was performed using G*Power version 3.1.9.6 for MAC OS.

15. Recruitment: Patients will be recruited by A.K. from outpatient clinic of conservative dentistry department in Faculty of Dentistry, Cairo University. Eligible patients will then be recruited to fulfill the eligibility criteria according to participant timeline.

B) Assignment of interventions 16. Allocation:

16a. Randomization: M.S. will perform simple randomization by generating numbers from 1 to 50, divided into two groups denoting letter A and B. Randomization will be done using random Sequence Generator, Randomness and Integrity Services Ltd (https://www.random.org/).

16b. Allocation concealment mechanism: The allocation sequence will be kept with the contributor (M.S.) in sealed tight envelopes concealed from the primary investigator. The principal investigator (A.K.) will know the allocation of the consented participant just before starting the operative procedures.

16c. Implementation Sequence generation and allocation concealment will be implemented by M.S.

17. Masking/blinding: The participants, assessors and statistician (A.Z. and S.H.) will be blinded to the material assignment, while the operator will not be due to the difference in restorative material presentation and its application protocol.

C) Data collection, management, and analysis:

18. Data collection methods

1. Baseline data collection: For every patient, medical and dental history will be taken. Examination charts will be filled by A.K.
2. Outcome data collection: Modified USPHS criteria for dental restoration will be evaluated by two assessors (A.Z. & S.H.) at baseline, after 6 and 12 months, if both assessors differ in score, they will discuss.

   19. Data management: All paper sheets that are concerned with the personal or outcome data will be stored in locked cabinet and in the computer. The excel sheets of the patient's data will be stored on a computer with a password only known to M.S. to prevent unauthorized access to data and double data entry.

   20. Statistical methods: Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 25 (SPSS Inc., Chicago, IL). Categorical data will be described as absolute risk for each intervention independently and relative risk when comparing both interventions. Comparisons between categorical variables will be performed using the chi-square test and Kruskal Wallis will be used to test the interaction of variables. Continuous data will be described using mean and standard deviation. Comparison between continuous data will be performed using T-test and ANOVA to test the interaction of variables. A p-value less than or equal to 0.05 will be considered statistically significant and all tests were two-tailed.

   D) Data monitoring:

   21. Monitoring Supervisors A.Z. and S.H. will monitor this study. Their role is to monitor any risk of bias from participants, operator or assessors, monitor blinding of the assessors and monitor patient safety and outstanding benefits or harms.

   22. Harms Operator A.K. should inform participants about the possible harms (pain, loss of restoration, leakage and fracture of restorations) if present. Participants are allowed to contact the operator at any moment through telephone. For assessment radiograph, inspection, percussion and sensitivity tests will be performed. The data will be reported to the main supervisor and managed through removal of restoration, alleviation of pain and replacement with control restoration.

   23. Audit In this trial auditing will be done by the supervisors A.Z. and S.H. to assure the quality of the research methods, preventive techniques and interventions.

   IV. Ethics and dissemination

   24. Research ethics approval Application forms for carrying out the clinical trial, checklist, and informed consent of Research Ethics Committee (REC) Faculty of Dentistry, Cairo University will be retrieved and filled, then will be delivered for (REC) committee for approval; this is done to prevent any ethical problems during the study or any harm for any of the participants.

   25. Protocol amendments If a new protocol is to be implemented, a protocol amendment will be submitted. This will include a new version of the protocol, and a brief explanation of the differences compared to previous versions. Additionally, any changes to the existing protocol that impact the safety of participants, scope of investigation, or scientific quality of the trial will be communicated through an amendment with a brief explanation of the modifications. Furthermore, if a new author is to be added to facilitate the study, an amendment will be submitted that includes the investigator's credentials and qualifications, aiming to prevent ghost authorship.

   26. Informed consent The principal investigator A.K. will be tasked with obtaining and signing the informed consents on the day of enrollment. The model of the Research Ethics Committee (REC) of the Faculty of Dentistry, Cairo University, will be utilized throughout this clinical trial.

   27. Confidentiality Name and personal data of the participants will not appear on the protocol form and will be maintained secured for 5 years after the trial. This is done for the protection of participants' privacy and civil rights.

   28. Declaration of interest There is no conflict of interest, no funding or material supply from any parties. The protocol is self-funded by the principal investigator.

   29. Access to data Access to final data will be allowed to the operator and main supervisor and co supervisors of the study who are not involved in the assessment of the outcome 30. Post-trial care Patients will be followed up after restoration to ensure oral hygiene measures. When there is any evidence of restoration failure, patients will be treated by immediate restoration removal and direct composite restoration will be placed.

   31. Dissemination policy Full protocol will be published online in Clinicaltrials.gov to avoid repetition and keep the integrity of the research work. Thesis will be discussed and defended in front of a judgment committee. The study will be published to report the results of this clinical trial.

   V. Appendices 32. Appendix Appendix 1: MBU acceptance. Appendix 2: Clinical trials registration. Appendix 3: Informed consent. Appendix 4: human ethics application form. VII. Statement of originality

   33. Statement of originality I declare this research submitted to Faculty of Dentistry, Cairo University is considered my original work done under the supervision and guidance of Professor Dr. Ahmed Al Zohairy, Prof. Dr. Shereen Hafez. All the information and data in this research are authentic, and all sources used are fully referenced. This research has never been submitted before to anyone or anywhere; not to any other universities or institutions.

ELIGIBILITY:
Inclusion Criteria:

For Participants:

* Age: 18-60 years.
* Males or females.
* Participants with endodontically treated molar teeth. Lower molars indicated for onlay (one or two missing cusps)
* Patients with at least 20 teeth under occlusion.
* Good oral hygiene.
* Co-operative patients approving to participate in the trial.
* Have sufficient cognitive ability to understand consent procedures.

For Teeth:

Badly destructed endodontically treated molars teeth indicated for cuspal total cuspal coverage (Overlay restoration)

* No signs or symptoms after endodontic treatment.
* No signs of clinical mobility.
* Teeth with healthy periodontium.

Exclusion Criteria:

For Participants:

* Participants with parafunctional habits or bruxism.
* Participants with systemic diseases or disabilities that may affect participation.
* Heavy smoking.
* Pregnancy.
* Lack of compliance.
* Severe or active periodontal disease.
* Cognitive impairment for teeth:
* Periapical pathosis indicating failure in endodontic treatment.
* Vital teeth.
* Signs of pathological wear.
* Severe periodontal affection or tooth indicated for extraction.
* Signs of Vertical root fracture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Restoration Integrity, Fracture | measurements will be taken Immediate Post restorative, 6 month, 12 month & 18 month follow ups
  Primary outcome will be measured using modified USPHS Criteria with A,B & C grades A: No evidence of restoration fracture. B: Minor chipping of restoration prone to repair. C: Severe chipping or bulk fracture beyond repair.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic, Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nam, N.E., Hwangbo, N.K., Kim, J.E., 2024. Effects of surface glazing on the mechanical and biological properties of 3D printed permanent dental resin materials. J. Prosthodont. Res. 68, 273-282. https://doi.org/10.2186/jpr.JPR_D_22_00261 Özden, Y., Altınok Uygun, L., 2025. Effects of postcuring times on the trueness of 3D -printed dental inlays made with permanent resins. Clin. Oral Investig. 29. https://doi.org/10.1007/s00784-025-06319-z
- [Background] Mudhaffer, S., Haider, J., Satterthwaite, J., Silikas, N., 2025. Effects of print orientation and artificial aging on the flexural strength and flexural modulus of 3D printed restorative resin materials.Manchester,UK.https://doi.org/ns.org/licenses/by/4.0/).https://doi.org/10.1016/j.prosdent.2024.08.008
- [Background] Metin, D.S., Schmidt, F., Beuer, F., Prause, E., Ashurko, I., Sarmadi, B.S., Unkovskiy, A., 2024. Accuracy of the intaglio surface of 3D-printed hybrid resin-ceramic crowns, veneers and table-tops: An in vitro study. J. Dent. 144. https://doi.org/10.1016/j.jdent.2024.104960
- [Background] Lim, B., Kim, D., Song, J.S., Kim, S., Kim, H., Shin, Y., 2024. Influence of Post-Curing in Nitrogen-Saturated Condition on the Degree of Conversion and Color Stability of 3D-Printed Resin Crowns. Dent. J. (Basel). 12. https://doi.org/10.3390/dj12030068